CLINICAL TRIAL: NCT00248794
Title: The Effects of Cognitive Rehabilitation on Function in Schizophrenia
Brief Title: Cognitive Rehabilitation in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: O3251-R; 00471 (Other: VA CT)
Record Dates: First submitted 2005-11-02; First posted 2005-11-04 (Estimated); Results first posted 2016-04-14 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-04

CONDITIONS: Cognitive Impairment; Schizophrenia
Keywords: Cognitive Impairment; Rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction; Schizophrenia | interventions — secoisolariciresinol; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CRT + Skills Training (Experimental): The intervention is call Cognitive Remediation Therapy (CRT) with a skill development group. Participants receive 15 weeks of cognitive training (with intake, 15 and 30 week assessment). This intervention is reliant upon didactic exchanges between trainer and participant, minimizing error, and behavioral modeling with the goal of developing better meta-cognitive skills. Procedures include paper and pencil activities (memory, planning and cognitive flexibility training) which are organized by difficulty. Sessions are organized to have a discussion between the trainer and the participant about the task and strategies, trainer modeling with articulation of strategy a participant attempts the task, talking aloud the steps, and finally the participant practices the task covertly. The trainer has the role of "error catcher and model." All subjects randomized to this condition also are receiving the weekly skills group (SDG)offered to participants in all experimental conditions.
  Interventions: Behavioral: Cognitive Rehabilitation Therapy (CRT) + Skill Training (SDG)
- ICBCR and Skills Training (Experimental): This intervention is Individualized Computer Based Cognitive Remediation (ICBCR) and skills development group (SDG). Participants receive 15 weeks of computerized training (with intake, 15 and 30 week assessments). This intervention relies upon intense, frequent, repetition of tasks being made incrementally more challenging. Computer tasks are organized so that the initial trials are easily completed and more challenging levels are then attempted. Parameters such as duration of task, task speed, and intra-task variables all be are manipulated. A trainer will be present at each session to help set up the computer tasks and answer questions. Besides the first two sessions that will be orientation sessions, the trainer has little involvement during the training sessions. The role of the trainer is to help organize, support, and provide feedback to each participant. All subjects randomized to this condition also are receiving the weekly skills group (SDG).
  Interventions: Behavioral: Individual Computer Based Cognitive Rehabilitation (ICBCR) and Skills Training (SDG)
- Skills Group Control (Experimental): The control intervention is call the skills development group (SDG) and is augmented with up to five individual contacts with research staff. The Skills Group (SDG) control is standard care group which will receive 15 weeks of the skills development group (SDG) similar to that offered as a clinical service at the VA Medical Center. During the 15 weeks participants will attend 1.5 hours of skills group per week. The 15 sessions will include skills training related to: a) cooking and food preparation, b) negotiating the local transportation system, c) shopping, and d) planning leisure activities. The training activities are a blend of didactic learning, modeling and finally in vivo practice. Participants in this group will also be offered up to five weekly contacts with staff to balance out factors related to meeting with staff in the other conditions.
  Interventions: Behavioral: Skills Group (SDG)

INTERVENTIONS:
Behavioral: Cognitive Rehabilitation Therapy (CRT) + Skill Training (SDG) — CRT is a one on one cognitive skills training and Skill training is a group intervention to develop concrete skills of daily living.
  Arms: CRT + Skills Training
Behavioral: Individual Computer Based Cognitive Rehabilitation (ICBCR) and Skills Training (SDG) — ICBCR is a computerized cognitive skills training program and Skill training is a group intervention to develop concrete skills of daily living.
  Arms: ICBCR and Skills Training
Behavioral: Skills Group (SDG) — Skill training is a group intervention to develop concrete skills of daily living. This is augmented with the opportunity to receive up to 5 hours of individual staff contact.
  Other Names: Standard care
  Arms: Skills Group Control

SUMMARY:
The study will investigate the viability of two cognitive rehabilitation strategies to improve functional outcomes for people with schizophrenia. Many people with schizophrenia experience impairments in cognitive function which limit their abilities. These impairments have been shown to precede the onset of illness and represent a vulnerability factor which is exacerbated by emerging psychotic symptoms. These impairments affect a range of functional domains including symptom severity, work function, symptom management, treatment, and overall quality of life. Recognizing the link between cognitive impairment and function, a few clinicals and researchers have attempted to remediate cognitive impairments by providing cognitive retraining programs similar to those used in traumatic brain injured patients or adaptive skills training. Cognitive retraining involves repetitive exercises to increase elemental cognitive functions including memory, attention, psychomotor speed, planning, and cognitive flexibility. Adaptive skill training involves didactic group exercises in social skills, activities of daily living, and symptom management. Each approach has demonstrated some rehabilitation benefits. This study will investigate the effectiveness of a combination of these two approaches on outcomes in schizophrenia.

DETAILED DESCRIPTION:
Objective: Many people with schizophrenia experience impairments in cognitive function which limit their abilities. These impairments affect a range of functional domains including symptom severity, work function, symptom management, treatment, and overall quality of life. Recognizing the link between cognitive impairment and function, a few clinicians and researchers have attempted to remediate cognitive impairments by providing cognitive retraining programs similar to those used in traumatic brain injured patients or adaptive skills training. Cognitive retraining involves repetitive exercises to increase elemental cognitive functions including memory, attention, psychomotor speed, planning, and cognitive flexibility. Adaptive skill training involves didactic group exercises in social skills, activities of daily living, and symptom management. This study investigates the effectiveness of a combination of these two approaches on outcomes in schizophrenia. This will be a three group randomized clinical trial investigating the effects of cognitive rehabilitation on outcomes ranging from proximal (training tasks performance and neuropsychological test performance), to more distal outcomes (treatment group performance and quality of life ratings). We believe that the cognitive augmentation will have significant impact on training task and neuro-psychological test performance and attenuated, but significant effect on performance in the treatment groups. Finally, we hypothesize that the combination of adaptive training and cognitive rehabilitation will have measurable impact on the most distal outcomes such as daily living skills and quality of life. Method: One hundred (100) individuals will be invited to participate in a 30-week program. After informed consent is obtained and diagnosis established, participants will receive an extensive assessment of neuropsychological, psychological and psychosocial functioning. Participants will be randomly assigned to one of three conditions using a stratified procedure based on cognitive test performance (this will ensure that there are similar numbers of severely and less severely impaired participants in each condition). The three conditions will be: (1) a usual care control group which is the Life Skills Development Group (LSDG), (2) Individualized computer based cognitive rehabilitation (ICBCR) augmenting the LSDG; and (3) Cognitive Remediation Therapy (CRT) with LSDG. Participants will be compared on: (1) LSDG performance, (2) neuropsychological test performance and (3) psychosocial functioning. Attendance in groups and remediation sessions will be compensated at a rate of $5 per session. The key questions t be answered are which Cognitive Rehabilitation strategy is more effective at improving cognitive function? Does Cognitive Rehabilitation produce better performance in the Life Skills Development Group (LSDG)? Does Life Skills Development Group augmented by Cognitive Rehabilitation produce better psychosocial outcomes than the standard care control group?

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia or schizoaffective disorder. Between the ages of 18-65. Stable medication regime (no changes in last 30 days)Minimum of 30 days since last hospitalization. No hx of TBI

Exclusion Criteria:

* Current Substance abuse, no comorbid neurological disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2004-06; Primary Completion 2008-12 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Bryson, Principal Investigator — VA Connecticut Health Care System (West Haven)
Locations (1):
- VA Connecticut Health Care System (West Haven), West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Data to be written up in peer review journal and possibly presented at regional and national conferences, but there is no plan to de-identify and share

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans with schizophrenia or schizoaffective disorder who met the following inclusion were recruited between 2004 and 2008.
Groups:
- CRT + Skills Training: Cognitive Remediation therapy+ skills training
  Participants received up to 5 hours of CRT and weekly skills training group
- ICBCR and Skills Training: Individualized Computer Based Cognitive Remediation
  Participants received up to 5 hours of ICBRC and weekly skills group
- Skills Group Control: Participants received weekly skills group + up to five individual contacts with research staff without active cognitive training
Period: Overall Study
Arm/Group | CRT + Skills Training | ICBCR and Skills Training | Skills Group Control
Started | 25 | 24 | 10
Completed | 19 | 16 | 7
Not Completed | 6 | 8 | 3
Not completed — Lost to Follow-up | 6 | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- CRT +Skills Group: Participants receive upto 5 hours of CRT and weekly skills training group for 15 weeks
- ICBCR + Skills Group: Participants receive upto 5 hours of ICBCR and weekly skills training group for 15 weeks
- Skills Group Only: Participants receive upto 5 hours of generic staff contact and weekly skills training group for 15 weeks
- Total: Total of all reporting groups
Arm/Group | CRT +Skills Group | ICBCR + Skills Group | Skills Group Only | Total
Number analyzed (Participants) | 25 | 24 | 10 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (6.7) | 47.6 (8.1) | 48.1 (6.9) | 47.8 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 1 | 9
  Male | 21 | 20 | 9 | 50
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 10 | 59

OUTCOME MEASURES:

1. Primary Outcome: Wisconsin Card Sort Percent Perseverative Errors (Standard Score)
Description: This is a measure of cognitive flexibility and the ability to shift set in the face of a changing reinforcement. The measure reflects "density" of perseverative errors in relation to the overall test performance. It is computed by calculating the ration of perseverative errors to trials administered and multiplied by 100. Then the percentage score is translate using the available Standard Score Tables provided in the manual and converted to a standard score with a mean of 100, a maximum of 145 and a minimum of 55, with higher Standard Scores indicating better performance.
Time Frame: 16 weeks after intake
Measure: Mean (Standard Deviation); unit: standard score units
Groups:
- CRT + Skills Training: Cognitive Remediation therapy-Up to 5 hours of one on one cognitive remediation using CRT. All subjects randomized to this condition also are receiving the weekly skills group.
  Cognitive rehabilitation (CRT and ICBCR): CRT is a one on one cognitive skills training method while ICBCR is a computer-based methods to improve cognitive abilities
- ICBCR and Skills Training: Individualized Computer Based Cognitive Remediation-Up to 5 hours of of computer based cognitive remediation (ICBCR). All subjects randomized to this condition also are receiving the weekly skills group.
  Cognitive rehabilitation (CRT and ICBCR): CRT is a one on one cognitive skills training method while ICBCR is a computer-based methods to improve cognitive abilities
- Skills Group Control: Life skills group + up to five individual contacts with research staff without active cognitive training
Arm/Group | CRT + Skills Training | ICBCR and Skills Training | Skills Group Control
Number analyzed (Participants) | 25 | 24 | 10
standard score units | 87.54 (4.04) | 87.88 (3.98) | 91.80 (6.30)
Statistical Analysis 1: Comparison: CRT + Skills Training vs ICBCR and Skills Training vs Skills Group Control; Test type: Superiority or Other; p < .97, ANOVA

2. Primary Outcome: Bell Lysaker Emotion Recognition Test
Description: 21 Item audio-visual task that measures the ability to recognize affective states in others. Affective states presented include: Happiness, Sadness, Surprise, Disgust, Fear, Anger and No Emotion. The instrument is scored for total correct responses with scores ranging from 0 to 21 with higher scores indicate better overall performance.
Time Frame: 16 weeks from intake
Population: Two way ANOVA using baseline and completion of intervention data
Measure: Mean (Standard Deviation); unit: total correct
Arm/Group | CRT + Skills Training | ICBCR and Skills Training | Skills Group Control
Number analyzed (Participants) | 25 | 24 | 10
total correct | 14.17 (.74) | 13.40 (.73) | 14.50 (1.15)
Statistical Analysis 1: Comparison: CRT + Skills Training vs Skills Group Control; Test type: Superiority or Other; p = .77, ANOVA

3. Primary Outcome: Continuous Performance Task X/A Version
Description: CPT relative X/A Percentage. This is a task-oriented computerized assessment of attention-related problems. This variable measures the relative sustained attention, and vigilance over the time of the task. Raw performance is standardize using available age and education norms yielding a Standardized Score with a mean of 100. Maximum Standard score is 145 and the minimum is 55 with higher scores reflect better performance.
Time Frame: 16 weeks after intake assessment
Measure: Mean (Standard Deviation); unit: units on a scale (standardized units)
Arm/Group | CRT + Skills Training | ICBCR and Skills Training | Skills Group Control
Number analyzed (Participants) | 24 | 25 | 10
units on a scale (standardized units) | 91.31 (3.55) | 92.65 (3.48) | 92.17 (5.50)

4. Primary Outcome: Hopkins Verbal Learning Test- Total Recall Variable
Description: This is measure of verbal learning and memory for immediate recall. Respondents are read a list of 12 items and asked to repeat once the last item is given. The list if given 3 times. Each time all items are recorded giving a total score ranging from 0 to 36. The score is converted to T-scores (mean of 50 and sd of 10) using the norms in the manual. The data reported are that in T-Scores with higher scores indicating better functioning.
Time Frame: 16 weeks post intake assessment
Measure: Mean (Standard Deviation); unit: units on a scale (T-scores)
Groups:
- CRT + Skills Training: Participants receive upto 5 hours of CRT and weekly skills training group for 15 weeks
- ICBCR and Skills Training: Participants receive upto 5 hours of ICBCR and weekly skills training group for 15 weeks
- Skills Group Control: Participants receive upto 5 hours of generic staff contact and weekly skills training group for 15 weeks
Arm/Group | CRT + Skills Training | ICBCR and Skills Training | Skills Group Control
Number analyzed (Participants) | 24 | 25 | 10
units on a scale (T-scores) | 36.33 (2.19) | 32.56 (2.14) | 32.90 (3.39)

5. Primary Outcome: Independent Living Skills Survey
Description: Independent Living Skills Survey is a 103 items that assess 12 areas of skills; personal hygiene (6 items), appearance and care of clothing (12 items), care of personal possessions and living space (9 items), food preparation (9 items), care of one's own health and safety (10 items), money management (10 items), transportation (7 items), leisure and recreational activities (13 items), job seeking (6 items), job maintenance (3 items), eating behaviors (9 items), and social interactions (9 items). The items describe relatively specific skills such as "washes hair twice a week," and informants indicate how frequently an individual has performed each skill within the past month. The responses are yes (1 point) no (0 points). Scores reports are the average #of yes items/number of total items. Higher scores indicating better functioning.
Time Frame: 16 weeks after intake
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CRT + Skills Training | ICBCR and Skills Training | Skills Group Control
Number analyzed (Participants) | 24 | 25 | 10
units on a scale | .73 (.02) | .73 (.02) | .77 (.04)

ADVERSE EVENTS:
Time Frame: 2004-2008
Groups:
- CRT+Skills Group: Cognitive Remediation therapy-Up to 5 hours of one on one cognitive remediation using CRT. All subjects randomized to this condition also are receiving the weekly skills group.
  Cognitive rehabilitation (CRT and ICBCR): CRT is a one on one cognitive skills training method while ICBCR is a computer-based methods to improve cognitive abilities
- ICBCR + Skills Group: Individualized Computer Based Cognitive Remediation-Up to 5 hours of of computer based cognitive remediation (ICBCR). All subjects randomized to this condition also are receiving the weekly skills group.
  Cognitive rehabilitation (CRT and ICBCR): CRT is a one on one cognitive skills training method while ICBCR is a computer-based methods to improve cognitive abilities
- Skills Group + Generic Contact: Life skills group + up to five individual contacts with research staff without active cognitive training
Arm/Group | CRT+Skills Group | ICBCR + Skills Group | Skills Group + Generic Contact
Serious Adverse Events (participants affected / at risk) | 2/25 | 1/24 | 1/10
Other Adverse Events (participants affected / at risk) | 6/25 | 7/24 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT+Skills Group (N=25) | ICBCR + Skills Group (N=24) | Skills Group + Generic Contact (N=10)
increase in psychiatric symptoms (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) — subject had increase in psychiatric symptoms requiring hospitalization
Cardiac event (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Subject had cardiac event and had to be hospitalized from home not while engaged in the intervention, but during the intervention period
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT+Skills Group (N=25) | ICBCR + Skills Group (N=24) | Skills Group + Generic Contact (N=10)
sought non psychiatric medical attention in ER (General disorders) | 4 (7) | 5 (9) | 2 (4)
Went to Psych ER but was not hospitalized (Psychiatric disorders) | 2 (4) | 2 (5) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes